CLINICAL TRIAL: NCT03595475
Title: Prodromal Markers of α-synucleinopathy Neurodegeneration in the First-degree Relatives of Patients With Psychiatric Disorders Comorbid With REM Sleep Behavior Disorder
Brief Title: Prodromal Markers of First-degree Relatives of Patients With Psychiatric Disorders Comorbid With RBD
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Wing Yun Kwok, Professor, Chinese University of Hong Kong
Other Study IDs: RGC14172917
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: REM Sleep Behavior Disorder
Keywords: Prodromal markers; Psychiatric disorders; α-synucleinopathy; Family study
MeSH Terms: conditions — REM Sleep Behavior Disorder; Mental Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample will be taken for genetic study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Psychiatric RBD cases: 1. Presence of REM sleep without atonia;
  2. At least one of the followings is present: i). Dream enactment behaviors, SRIs, potentially injurious or disruptive behaviors by history; ii). Abnormal REM sleep behaviors documented during v-PSG monitoring;
  3. Absence of electroencephalogram (EEG) epileptiform activity during REM sleep unless RBD can be clearly distinguished from any concurrent REM sleep related seizure disorder;
  4. The sleep disturbance is not better explained by other sleep disorder (e.g., obstructive sleep apnea, medical or neurological disorder, mental disorder, medication use, or substance use disorder)
- Psychiatric control: 1. Age- and sex- matched with pRBD proband;
  2. Concurrent psychiatric illnesses according to the Mini International Neuropsychiatric Interview( M.I.N.I);
  3. Free of narcolepsy and other neurological diseases;
  4. Absence of any RBD features as based on REM sleep behavior disorder questionnaire (RBDQ-HK) and v-PSG; 5) Free of neurodegenerative diseases
- Healthy control: 1. Age- and sex- matched with pRBD proband;
  2. Without lifetime psychiatric disorder according to Mini International Neuropsychiatric Interview( M.I.N.I);
  3. Free of narcolepsy and other neurological diseases;
  4. Absence of any RBD features as based on RBDQ-HK and v-PSG;
  5. Free of neurodegenerative diseases

SUMMARY:
REM sleep behavior disorder (typical or 'idiopathic' RBD, iRBD) is a novel and distinct parasomnia characterized by recurrent dream enactment behaviours and polysomnographic features of loss of normal REM-sleep related muscle atonia, with a male predominance commonly occurring at the age of 60's. A majority of the patients with iRBD will eventually develop α-synucleinopathy (e.g., Parkinson's disease). On the other hand, growing evidence reveals a specific group of psychiatric patients demonstrating comparable clinical RBD features (pRBD) (e.g., abnormal REM-related electromyographic (EMG) activities) as found in typical iRBD, but with less male predominance occurring at the age of mid 40's to early 50's. Although recent findings from both cross-sectional and prospective studies have suggested that pRBD is likely to be a persistent parasomnia with close association with clinical and neuroimaging biomarkers related to neurodegeneration, the nosology of the development of RBD symptoms among patients with psychiatric disorders, notably major depressive disorder, remains unclear as to whether they are simply antidepressants related, or represent a part of the early phase of α-synucleinopathy neurodegeneration. Family studies on iRBD have confirmed a significant familial aggregation of iRBD with a higher rate of RBD cases and presence of prodromal neurodegenerative biomarkers (e.g. tonic EMG activity during REM sleep, constipation, and motor function impairments) of α-synucleinopathy neurodegeneration among first-degree relatives (FDRs) of patients with iRBD. Thus, the investigators propose this family study to examine the following hypotheses: 1) FDRs of patients with pRBD have a higher rate of RBD symptoms and its core features when compared to FDRs of controls with and without psychiatric disorders; 2) FDRs of pRBD are more likely to exhibit the features associated with prodromal markers of α-synucleinopathy neurodegeneration when compared with FDRs of controls with and without psychiatric disorders; 3) FDRs of patients with pRBD have a higher rate of α-synucleinopathy neurodegeneration when compared with FDRs of controls with and without psychiatric disorders. A total of 176 FDRs from each group (e.g., pRBD cases, psychiatric controls, and healthy controls) will be recruited to undergo a face-to-face clinical interview and a series of assessments on prodromal markers of Parkinson's diseases (as according to the International Parkinson and Movement Disorder Society research criteria) respectively.

All FDRs with possible RBD and a subset of FDRs without possible RBD will be invited to undergo one-night video-polysomnographic assessment to confirm the clinical diagnosis of RBD and to assess the abnormal REM-related EMG muscle activities.

DETAILED DESCRIPTION:
REM sleep behavior disorder (RBD) is a novel REM sleep parasomnia characterized by dream enacting behaviors and sleep-related injuries. Ample evidences have suggested that idiopathic RBD (iRBD) is a precursor of α-synucleinopathy neurodegeneration (e.g. Parkinson's disease, PD) in which dopamine dysfunction is one of the core pathophysiologies. In recent decade, our group has identified a cohort of patients with psychiatric disorders (mainly major depressive disorder, MDD) comorbid with RBD (pRBD). While there was a postulation that RBD symptoms in this psychiatric population may simply be side effects of antidepressant medication (by enhancing REM-sleep related muscle activity), accumulating evidence from case-control and prospective cohort studies suggested that pRBD is only partially explained by antidepressant usage and is better considered as a variant of typical iRBD in terms of comparable clinical presentation with typical iRBD and its close association with neurodegenerative markers. Nonetheless, more evidence is needed to substantiate that pRBD is a distinct diagnostic entity rather than a symptom secondary to antidepressant use. In this study, the investigators will employ genetic epidemiology approach to: 1) determine the familial genetic contribution; 2) search for biomarkers and endophenotypes; and 3) validate the diagnostic entity of a disease.

This proposed study will enrich the limited scientific literature of the potential pathogenesis of pRBD and its relationship with α-synucleinopathy. In addition, the understanding of psychiatric disorders, notably MDD, is often limited by its heterogeneity. Our proposed study will, by determining the familial aggregation of pRBD, help us to identify certain subtype of the psychiatric populations who may likely harbour an underlying neurodegenerative basis. By using a family study design, a number of important aspects with regard to the pathogenesis of pRBD will be answered. First, if first-degree relatives (FDRs) of patients with pRBD have a higher rate of possible RBD or clinical diagnosis of RBD (as confirmed by video-polysomnography) as well as the presence of neurodegenerative diseases when compared with FDRs of controls, it will substantiate the argument that pRBD is not merely a side effect of antidepressants but rather harbouring a familial and genetic predisposition to RBD and, ultimately α-synucleinopathy neurodegeneration. Second, the determination of biomarkers of neurodegeneration among unaffected FDRs of patients with pRBD will also help to identify high-risk individuals for clinical intervention and prevention. Third, the calculation of heritability will help to delineate to which extent the additive genetic contribution is responsible for the variance of pRBD phenotypes. Finally, the findings from this proposed study will be compared with our on-going family study of typical iRBD to determine the extent to which iRBD and pRBD are similar or different to each other in terms of genetic and familial associations.

In this proposed study, the investigators hypothesize that:

1. FDRs of patients with pRBD have a higher rate of RBD symptoms and its core features compared with FDRs of controls;
2. The unaffected FDRs of patients with pRBD are more likely to exhibit the features associated with prodromal markers of Parkinson's disease compared with FDRs of controls;
3. FDRs of patients with pRBD have a higher rate of Parkinson's disease (and other α-synucleinopathy neurodegeneration) compared with FDRs of controls.

ELIGIBILITY:
Inclusion Criteria:

* Age- and sex- matched with pRBD proband;
* Without lifetime psychiatric disorder according to Structural Clinical Interview for DSM-IV Disorders (SCID);
* Free of narcolepsy and other neurological diseases;
* Absence of any RBD features as based on RBDQ-HK and v-PSG;
* free of neurodegenerative diseases.

Exclusion Criteria:

* Not Chinese or aged under 40 years old;
* Refuse to participate in this study;
* without a biological relationship with proband.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, we will employ a combination of family history (proxy report for unavailable/inaccessible subjects) and study (face-to face interview, clinical and sleep study) method in determining the familial aggregation of pRBD. The flowchart of subject recruitments is presented in Figure 1. The study subjects are the FDRs of pRBD cases, psychiatric controls and healthy controls. As previous studies have suggested that depression is a significant risk factor of development of Parkinson's Disease, we will include two control groups. First, those FDRs of patients with psychiatric disorders in addition to the FDRs of healthy controls (free of depression and RBD), in consideration of the potential associations of proband's psychiatric disorders with prodromal markers of Parkinson's Disease in the FDRs.
Sampling Method: Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of possible REM Sleep Behavior Disorder | 17 months
  The prevalence of possible REM Sleep Behavior Disorder based on the self-reported/proxy-reported REM Sleep Behavior Disorder symptoms in REM Sleep Behavior Disorder Questionnaire-HK among First Degree Relatives,

SECONDARY OUTCOMES:
Percentage of REM-related EMG activity | 17 months
  The mean differences in the percentage of REM-related EMG activity among First Degree Relatives in different groups
Weighted prevalence of Polysomnography confirmed REM Sleep Behavior Disorder | 17 months
  Prevalence of Polysomnography confirmed REM Sleep Behavior Disorder according to ICSD-3 criteria among First Degree Relatives in different groups
Recurrence risk of Parkinson's disease | 17 months
  Risk of Parkinson's disease and other α-synucleinopathy neurodegeneration based on family history report and face-to-face interview among First Degree Relatives in different groups

CONTACTS AND LOCATIONS:
Overall Officials: Yun Kwok Wing, Professor, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - The Chinese University of Hong Kong, Hong Kong
  - Shatin Hospital, Shatin

IPD SHARING:
Plan to Share IPD: Undecided
In this stage, the investigators didn't decide which information of IPD will share with other researchers

REFERENCES:
- [Derived] Wang J, Lam SP, Huang B, Liu Y, Zhang J, Yu MWM, Tsang JCC, Zhou L, Chau SWH, Chan NY, Chan JWY, Schenck CH, Li SX, Mok VCT, Ma KKY, Chan AYY, Wing YK. Familial alpha-synucleinopathy spectrum features in patients with psychiatric REM sleep behaviour disorder. J Neurol Neurosurg Psychiatry. 2023 Nov;94(11):893-903. doi: 10.1136/jnnp-2022-330922. Epub 2023 Jun 30. PMID 37399287